CLINICAL TRIAL: NCT00349440
Title: Efficacy of Topical Cyclosporine Ophthalmic Emulsion for the Prevention and Treatment of Dry Eye Symptoms Following LASIK or Photorefractive Keratectomy
Brief Title: Efficacy of Cyclosporine for the Prevention and Treatment of Dry Eye Symptoms Following LASIK or Photorefractive Keratectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Karl Stonecipher, MD, Southeastern Laser and Refractive Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1121
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Cyclosporine, Refresh Plus
- 2 (Placebo Comparator)
  Interventions: Drug: Cyclosporine, Refresh Plus

INTERVENTIONS:
Drug: Cyclosporine, Refresh Plus — Cyclosporine 0.4ml (in the eye) on for 3 months instill one drop in randomized eye twice daily.
  Refresh Plus 0.4ml (in the eye) on for 3 months instill one drop in randomized eye twice daily.

SUMMARY:
The purpose of this study is to evaluate the effect of topical cyclosporine ophthalmic solution 0.05% (Restasis, Allergan) on the signs and symptoms of dry eye in patients undergoing LASIK or photorefractive keratectomy (PRK).

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 years old
* Mild-moderate symptoms of dry eye prior to surgery
* Scheduled to undergo bilateral LASIK or PRK
* Likely to complete all study visits and able to provide informed consent

Exclusion Criteria:

* Prior use of topical cyclosporine within the last 1 year
* Known contraindications to any study medication or ingredients
* Female of child bearing potential not using reliable methods of birth control, or pregnant or lactating females.
* Ocular disorders
* Active ocular diseases or uncontrolled systemic disease
* Active ocular allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Dry Eye Symptoms | 1.5 years

SECONDARY OUTCOMES:
Dry eye signs | 1.5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Karl Stonecipher, MD, Principal Investigator — Southeastern Laser and Refractive Surgery
Locations (1):
- Southeastern Laser and Refractive Surgery, Greensboro, North Carolina, United States